CLINICAL TRIAL: NCT06196684
Title: Early Safety and Clinical Efficacy of Mitral Allografts in Patients With Primary Tricuspid Valve Disease Scheduled for Tricuspid Valve Replacement
Brief Title: Early Safety and Clinical Efficacy of Mitral Allograft in Tricuspid Surgery
Acronym: ESEMATS
Status: Active, not recruiting | Type: Observational
Sponsor: Chelyabinsk Regional Clinical Hospital (Other Government)
Responsible Party: Principal Investigator, Mikhail Nuzhdin, Director, Chelyabinsk Regional Clinical Hospital
Other Study IDs: 26122023
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Allografts; Tricuspid Valve Insufficiency
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with primary tricuspid valve insufficiency scheduled for tricuspid valve replacement
  Interventions: Procedure: Mitral allograft implantation

INTERVENTIONS:
Procedure: Mitral allograft implantation — Tricuspid valve replacement with mitral valve allograft

SUMMARY:
The aim of the study is to evaluate early safety and clinical efficacy of mitral allografts in tricuspid valve replacement for primary tricuspid valve diseases.

DETAILED DESCRIPTION:
Early safety (morbidity, mortality rate, freedom from any valve related complication) along with mid-term clinical efficacy ( mid-term survival, freedom from reoperation, repeat endocarditis and other valve related complication ) is going to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary tricuspid valve disease and/or tricuspid bioprosthetic failure scheduled for tricuspid valve intervention.
* Intraoperative findings suggested for tricuspid valve replacement rather than repair.

Exclusion Criteria:

* Pregnancy
* Confirmed active drug addiction
* Progressive HIV-infection
* HIV-infected patients with CD4-cells count less than 250
* Patients with secondary tricuspid valve pathology (left-sided valve disease)
* LV Ejection fraction less than 50%

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary tricuspid valve disease
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2026-09-29 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Mortality (all cause and valve-related) | 30-day period
  Estimate rate of mortality (all cause and valve-related)

SECONDARY OUTCOMES:
Neurologic events | 30-day period
  any neurological events in 30-day period
Bleeding and transfusions | 30 days
  Freedom from major bleeding events
Cardiac structural complications | 30 days
  any structural cardiac complication
Acute kidney injury | 30 days
  freedom from type 3-4 AKI
Allograft valve dysfunction | 30 days
  freedom from allograft valve stenosis or regurgitation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiac Surgery, Chelyabinsk, Chelyabinsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: No